CLINICAL TRIAL: NCT03337451
Title: Follow up Protocol to the Open Label Phase I/II Study OPN-305-106: A Prospective, Open Label Phase I/II Study to Assess the Safety and Efficacy of Cycles of Intravenously Infused Doses of OPN-305 in Second-line and Third-line Lower (Low and Intermediate-1) Risk Myelodysplastic Syndrome (MDS)
Brief Title: Follow up Protocol to the Phase I/II Study of OPN-305 in Second-line or Third-line Lower Lower Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Opsona Therapeutics Ltd. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other); Montefiore Medical Center (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPN-305-110
Record Dates: First submitted 2017-10-18; First posted 2017-11-09 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — tomaralimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OPN-305 (Experimental)
  Interventions: Drug: OPN-305

INTERVENTIONS:
Drug: OPN-305 — Patients will receive study drug every 4 weeks

SUMMARY:
This protocol is a follow-up for patients receiving continuation of OPN-305 monotherapy treatment or combination treatment with azacitidine after completion of the dose confirming, dose expansion and HMA naïve parts of the main study OPN-305-106.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the OPN-305-106 study
* Principal Investigator adjudicated efficacy response defined as either transfusion independence", "stable disease", "minor HI-E response" or "major HI-E response" and in the opinion of the Principal Investigator the patient may benefit from continued treatment with OPN-305 monotherapy or combination treatment with azacitidine.
* Provide written informed consent for the follow up protocol.

Exclusion Criteria:

* Refusal to provide written informed consent
* Withdrawal from the OPN-305-106 study prior to the final EOT visit
* Plan to be included into another interventional investigational study.
* Progression of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence and types of Serious Adverse events | monthly through study completion, an average of 18 months
monitor ongoing efficacy responses | monthly through study completion, an average of 18 months
  To monitor ongoing efficacy responses defined as "transfusion independence". Transfusion independence is defined as 56 consecutive days where no RBC transfusions are given

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Houston, Texas, United States